CLINICAL TRIAL: NCT03082365
Title: Prevalence of Oral Findings in Adult Patients With Chronic Kidney Disease '' Cross Sectional 2 "
Brief Title: Oral Findings in Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maryam Ahmed Essam Abdel Salam (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Maryam Ahmed Essam Abdel Salam, BDS internal resident at oral medicine department, Cairo University
Organization: Cairo University (Other)
Other Study IDs: renal_oral findings
Record Dates: First submitted 2017-03-12; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Oral Disease; Chronic Kidney Diseases
Keywords: oral findings or oral manifestations; pre-dialysis or end stage renal disease
MeSH Terms: conditions — Mouth Diseases; Renal Insufficiency, Chronic; Oral Manifestations; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- pre-dialysis
- end stage renal disease

SUMMARY:
The patients with chronic kidney disease suffer from many oral problems affecting the quality of life. The aim of our study is to assess their oral health to provide the proper management and increase their awareness

DETAILED DESCRIPTION:
The study will be held in the Nephrology units at the Kasr Al-Ainy Cairo university hospital.

The data collected through the questionnaire will be obtained through an interview between the investigator and the patient. Clinical examination will be performed for both oral (soft tissue) and dental (hard) tissue. For patients undergoing dialysis, examination will be performed before dialysis therapy Selection bias: will be minimized by enrolling the participants in the study in a consecutive order of the entering the clinic.

Non-respondent bias: will be minimized by explaining to the participants the aim of the study and their importance and role in the study.

Incomplete records: will be excluded from statistical analysis with reporting the cause of not completing the record.

Using a precision of 5, a design effect set at 1 with 90% CI (confidence interval), a total sample size of 250 pre-dialysis patients and 200 end stage renal disease patients will be sufficient. The sample size was calculated by Epi info software.The sample will be divided between two researchers; each researcher will have 50% of the whole sample to collect

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients >18 years old with a diagnosis of non-dialysis chronic kidney disease at stage 2, 3 and 4.
2. Adult patients >18 years old with a diagnosis of end stage renal disease "stage 5".
3. Recorded data of Glomerular Filtration Rate for every patient.
4. Recorded data for dialysis patients (HCV, platelets count, creatinine, blood urea nitrogen, urea level and partial thromboplastin time).

Exclusion Criteria:

1. Adult patients <18 years.
2. End stage renal disease undergoing peritoneal dialysis.
3. Patients not physically able to participate in oral examination.
4. Patients with kidney transplantation.
5. Patients undergoing renal dialysis for reasons other than chronic kidney disease, such as acute renal failure, accidents, trauma, snake poisoning

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A convenience sample of adult patients diagnosed with chronic kidney disease attending at the Nephrology units at El Kasr Al-Ainy Cairo University Hospital will be enrolled in the study in a consecutive order
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Primary Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Oral mucosal lesions | 15 minutes
  Clinical examination according to WHO guidelines

SECONDARY OUTCOMES:
Periodontal condition | 10 minutes
  Basic periodontal examination
Hepatitis C Virus at dialysis stage | 10 minutes
  HCV antibodies in patient blood

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gautam NR, Gautam NS, Rao TH, Koganti R, Agarwal R, Alamanda M. Effect of end-stage renal disease on oral health in patients undergoing renal dialysis: A cross-sectional study. J Int Soc Prev Community Dent. 2014 Sep;4(3):164-9. doi: 10.4103/2231-0762.142006. PMID 25374834